CLINICAL TRIAL: NCT05899257
Title: Effects of Brief Immersive Training on the Metacognitive Capacities and Self-knowledge of Young People
Brief Title: Immersive Training on Metacognitive Capacities of Young People
Acronym: VRtraining
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: European Union (Other); Universitat Autonoma de Barcelona (Other)
Responsible Party: Principal Investigator, Dr. Guillem Feixas, Full Professor, University of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VRT001
Record Dates: First submitted 2023-05-14; First posted 2023-06-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Self; Self-Perception; Self Esteem
Keywords: mentalization; self-knowledge; reflective function; virtual reality; self-identity; mental map; sense of identity

STUDY DESIGN:
Intervention Model Description: Single-group pre-post design with a one-month follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immersive Training using EYME-Explore Your Meanings (Experimental): Immersive training based on the RGT and EYME to improve the metacognitive abilities and self-knowledge of young people.
  Interventions: Behavioral: Immersive Training using EYME

INTERVENTIONS:
Behavioral: Immersive Training using EYME — Psychological assessment based on the RGT with EYME-Explore Your Meanings, a digital platform to explore the structure and content of personal identity with Virtual Reality.

SUMMARY:
Metacognitive abilities and self-knowledge are necessary for psychological maturation and good mental functioning of individuals. It is generally agreed that an adequate representation of oneself and others is essential to establish functional interpersonal relationships. These metacognitive abilities are not adequately developed in patients with various mental health problems, such as personality disorders, eating disorders, psychosis, and depression, and are associated with the severity of the pathology.

Self-awareness is a central element that begins to consolidate during adolescence. For that reason, the investigators aim to evaluate the effects of immersive training on the metacognitive abilities and self-knowledge of young people. Based on the repertory grid technique (RGT), our research team has developed a brief immersive training to enhance metacognitive abilities. This intervention facilitates the exploration of personal identity in a safe environment. Specifically, it is an immersion in the person's own world of meanings using Virtual Reality (VR), with the Explore Your Meanings (EYME) tool, a technological platform created to help mental health professionals to enhance the personal development and therapeutic change of their clients. Expected results include an increase in participants' self-concept clarity, metacognition, and reflective function as well as a deeper knowledge about their relationship with various aspects of self-knowledge and self-esteem.

DETAILED DESCRIPTION:
INTRODUCTION

Metacognitive abilities and self-knowledge are necessary for psychological maturation and good mental functioning of individuals. Self-knowledge is a central element in cognitive and personality development that begins to be structured during adolescence and evolves during youth and even later stages. It can be considered as the "mental map" or theory people use to construe themselves, and others based on their personal experiences. Self-knowledge consists of the schemas or constructs people use to interpret events, organize their responses and actions, and for anticipating the future. The variables that reflect metacognitive abilities and self-knowledge are diverse in the scientific literature. The investigators highlight the following:

1. Self-concept clarity is understood as the degree to which the contents of the person's self-concept are clearly defined, with certainty, with consistency, and are experienced as internally and temporally stable (Campbell et al., 1996).
2. Metacognition refers to the ability to identify, understand and reflect on one's own and others' mental states (e.g., thoughts, desires, emotions) (Pedone et al, 2017).
3. Reflective Function (RF) refers to the operationalization of the mental processes underlying mentalizing (Katznelson, 2014), which is defined as the ability to understand or interpret one's own and others' mental states, either implicitly or explicitly (Fonagy & Bateman, 2008).
4. Self-knowledge is a broad term used in several studies (e.g., Carapeto & Feixas, 2020) and is understood as the construction of one's personality characteristics in relation to the constructs they perceive in others and to their own "ideal self".
5. Self-esteem is a classic concept, often related to the previous terms, referring to the person's evaluation of their self and their capabilities.

Given that a good development of metacognitive capacities and self-knowledge is considered fundamental for the optimal functioning of individuals and society, the investigators consider the need to generate tools and/or interventions that can improve and enhance their development to be essential. In accordance, several approaches are considered. Personal Construct Theory (Kelly, 1955) focuses on the study of personal identity, understood as the core constructs of a person, and offers valid instruments to enhance metacognitive abilities and transformative self-knowledge. Based on the repertory grid technique (RGT), our research team has developed a brief immersive training to enhance the described metacognitive capacities.

This intervention allows participants to explore their personal identity in a safe environment. Specifically, it is an immersion in the person's own world of meanings through Virtual Reality (VR), with the Explore Your Meanings (EYME) tool, a technological platform created to help mental health professionals to enhance the personal development and therapeutic change of their clients.

OBJECTIVES

The general objective of this research is to evaluate the effects of immersive training based on RGT and EYME on the metacognitive abilities and self-knowledge of young participants. The specific objectives are:

1. To verify the hypothesis that such training increases participants' self-concept clarity, metacognition, reflective function, and self-esteem.
2. To identify the relationships between these variables and their relationship with indicators of self-knowledge (e.g., current self/ideal self-discrepancy; cognitive conflicts) derived from the RGT.
3. To explore the general characteristics of the contents and structure of self-knowledge in young participants.
4. To examine the relationship of gender and other sociodemographic variables with the level of metacognitive capacities and self-knowledge in young participants.

PROCEDURE. Participants will be contacted by posting an announcement on Internet forums and social networks, asking to those interested in participating to access an online survey. The survey will begin with the informed consent form. After reading and accepting the informed consent, participants will be presented with sociodemographic questions, such as age, sex, country, employment, and marital status as well as whether they have a record of severe mental illness or substance misuse in the last year. As part of this initial assessment, the following questionnaires will be administered: LS, SCC, MSAS, RFQ-8, RSE, CORE-OM, and DASS-21 (see Outcome Measures Section).

Among those completing the survey, eligible participants will be invited to attend in person the three-session intervention. In all these sessions, the CORE-SFB will be administered at the beginning of the session to detect possible suicidal ideation. If so, the researcher in charge will deal with this problem (proposing referral, contact with family, or call to specialized services) instead of continuing with the investigation.

First session: The researcher will explain to the participant the purpose of the three sessions, which consists of increasing self-knowledge to promote personal development and growth. The family and relational context of the participant and possible difficulties or issues of concern will be explored as well as the areas that he/she believes can be improved by increasing his/her self-knowledge. A self-characterization (Kelly, 1955; Feixas & Villegas, 2000) will be requested as a homework assignment (minimum one paragraph, maximum one page) to be handed in during the following session.

Second session: As part of the intervention, self-characterization will be briefly discussed and the RGT applied using the digital platform EYME. It begins with a computer-assisted interview where the constructs of the participant are elicited and applied by means of a 7-point visual scale to the most significant people in their interpersonal world, in addition to the "self now" and the "ideal self" (Feixas, Alabèrnia-Segura & García-Gutiérrez, 2022). Other elements of the self or other constructs that appear relevant from the first session or in the self-characterization can be included.

Third session: The results of the data analysis provided by EYME will be discussed in terms of self-definition, possible areas for improvement, and discrepancies between the current self, the ideal self, and others, as well as possible internal conflicts. The constructs and significant people are visualized in a 3D space visible on a computer screen, in which the participant has an immersive exploration using VR, offering a powerful and clarifying experience about the person's schemas and perceptions of self and others, also with respect to their ideal image. The dialogue with the researcher during and after the immersive experience is oriented towards facilitating the assimilation of the information provided and its analysis, which may include upward laddering from one of the relevant constructs of the person (Neimeyer, 1993). At the end of the session, the LS, SCC, MSAS, RFQ-8, RSE, and DASS-21 questionnaires will be administered.

Follow-up assessment: One month after the third session (placed two weeks after baseline), the CORE-OM, SCC, MSAS, RFQ-8, RSE, LS, and CRES-4 instruments will be administered online.

DATA ANALYSES. The statistical analysis will be carried out with Stata 16.1 (StataCorp LLC), and the reporting will be in accordance with the Statistical Analyses and Methods in the Published Literature (SAMPL) guidelines. Multivariate data normality distribution will be tested by the Mardia´s coefficients of skewness and kurtosis, and the univariate data normality distribution will be tested by the Shapiro-Wilk test. Overlap among variables will be examined with bivariate Spearman's correlations, and the collinearity by with the variance inflation factor (VIF).

A descriptive analysis of the sociodemographic and psychological variables will be performed. Multilevel linear mixed models of repeated measures will be conducted to assess the effect of the intervention, analyzing the pre- and post-scores of the outcome variables of SCC, MSAS, RFQ-8, and RSE, adjusted with the covariates of age, gender, and other sociodemographic variables. The method of estimation will be the Restricted Maximum Likelihood (REML), which is robust for moderate deviations of normality of continuous outcome variables. The adjustment of the model will be assessed with the Likelihood-Ratio test, the R2, the R2 adjusted, and the Bayesian Information Criteria (BIC). For all analyses, the significance level will be taken as 0.05, the confidence intervals will be calculated, and the effect size (Cohen's d) will be reported.

To achieve the second specific objective, correlations will be calculated between the variables related to the metacognitive abilities assessed with the SCC, MSAS, RFQ-8, RSE instruments, and the self-knowledge measures derived from the RGT. The inclusion of the CORE-OM will make it possible to assess the degree of change achieved with respect to psychological distress. Likewise, the application of CORE-SFB in each session will make it possible to evaluate the suicide risk and percentage of change session by session. With the DASS it will be possible to observe if there have been variations in the levels of anxiety, depression, and stress, although they are not expected to be high at the onset because it is a non-clinical sample.

A secondary analysis will be performed considering LSS as an outcome variable, in order to assess the evolution of a positive result, and its relationship with the other results will also be examined by means of a correlational analysis.

For the exploratory content analysis, two raters will code the constructs collected through the RGT, discuss disagreements found (if any), and perform a descriptive analysis. Inter-rater agreement will be calculated using the Kappa index.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between 18 and 29 years of age

Exclusion Criteria:

* Diagnosis of a mental disorder (current or in the last year)
* Current psychological or psychiatric treatment
* Suicidal ideation
* Insufficient level of competence to communicate in Spanish or English

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Self Concept Clarity after two weeks, and at one-month follow-up | SCCS will be administered at baseline, after two weeks, and at one-month follow-up.
  Self-concept clarity is assessed with the Self-Concept Clarity Scale (SCCS) created by Campbell et al. (1996) and adapted to Spanish by Feixas, et al (2023).
Change from baseline Metacognition after two weeks, and at one-month follow-up | MSAS will be administered at baseline, after two weeks, and at one-month follow-up.
  Metacognition will be assessed with the Metacognition Self-Assessment Scale (MSAS) created by Semerari et al. (2003) and adapted to Spanish by Feixas, et al. (2023).
Change from baseline Reflective Functioning after two weeks, and at one-month follow-up | Frame: RF will be administered at baseline, after two weeks, and at one-month follow-up.
  Reflective Functioning or mentalization will be assessed using the Reflective Functioning Questionnaire (RFQ-8) created by Fonagy et al. (2016) and adapted to Spanish by Ruiz-Parra et al (2023).

SECONDARY OUTCOMES:
Change from baseline Self-esteem after two weeks, and at one-month follow-up | RSE will be administered at baseline, after two weeks, and at one-month follow-up.
  Self-esteem will be assessed using the Rosenberg Self-Esteem Scale (RSE), a scale created by Rosenberg (1965) and adapted to Spanish by Martín-Albo et al. (2007) and Morejón et al. (2004).
Change from baseline Psychological distress, after one and two weeks, and at one-month follow-up | CORE-OM will be administered at baseline, after one and two weeks (using short forms version CORE-SFB), and at one-month follow-up.
  The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM; Evans et al, 2002), a 34-item self-report questionnaire, will be used for the assessment of subjective wellbeing, symptoms or problems, life functioning and risk. It has good psychometric properties (Trujillo et al, 2016) and it has been adapted into Spanish for free distribution (www.ub.edu/terdep/core). The short version (CORE-SFB) of 18 items will be used for session-to-session monitoring of the intervention process.
Change from baseline Depression, Anxiety and Stress, after two weeks and at one-month follow-up | DASS-21 will be administered at baseline, after two weeks, and at one-month follow-up.
  Depression, Anxiety and Stress Scales (DASS-21; Lovibond & Lovibond, 1995) is a 21-item version of the DASS and comprises 7 items for its three scales (depression, anxiety and stress), which are moderately correlated with each other. For Spanish speaking participants we will the Spanish adaptation (Bados, Solanas, & Andrés, 2005).
Change from Life Satisfaction after two weeks, and at one-month follow-up | LSS will be administered at baseline, after two weeks, and at one-month follow-up.
  The level of global satisfaction with life will be assessed with the Life Satisfaction Scale (LSS), which consists of a single item with a 10-point Likert scale response line.
Satisfaction with intervention | CRES-4 will be administered at the one-month follow-up.
  The degree of satisfaction with the intervention received is assessed with the Consumer Reports Effectiveness Scale (CRES-4; Feixas et al, 2012), which consists of four items.

OTHER OUTCOMES:
Self-knowledge | Self-knowledge assessment will be conducted after one week.
  Self-knowledge will be assessed with the RGT (Kelly, 1955; Feixas & Cornejo, 1996; Fransella, Bell & Bannister, 2004). The interview will be conducted with the assistance of the EYME platform. From the repertory grid data matrix, cognitive indices such as the current self - ideal self discrepancy, cognitive differentiation, polarization, presence and number of dilemmatic constructs, and implicative dilemmas will be obtained with the RECORD 6.0 program (Garcia-Gutierrez & Feixas, 2018; available at Internet: www.repertorygrid.net).

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Feixas, PhD, Principal Investigator — University of Barcelona
Locations (1):
- University of Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for all primary and secondary outcomes, after deidentification
Supporting Information: Study Protocol
Time Frame: Data will be available after six months of study completion
Access Criteria: Researchers who provide a methodologically sound proposal whose proposed use of the data has been approved by an independent review committee

REFERENCES:
- [Background] Bados, A., Solanas, A. y Andrés, R. (2005). Psychometric properties of the Spanish version of Depression, Anxiety and Stress Scales. Psicothema, 17, 679-683.
- [Background] Campbell, J. D., Trapnell, P. D., Heine, S. J., Katz, I. M., Lavellee, L. F., y Lehman, D. R. (1996). Self-concept clarity: Measurement, personality correlates, and cultural boundaries. Journal of Personality and Social Psychology, 70, 141-156
- [Background] Carapeto MJ, Feixas G. The Organization of Self-Knowledge in Adolescence: Some Contributions Using the Repertory Grid Technique. Eur J Investig Health Psychol Educ. 2020 Feb 5;10(1):408-423. doi: 10.3390/ejihpe10010031. PMID 34542494
- [Background] Evans C, Connell J, Barkham M, Margison F, McGrath G, Mellor-Clark J, Audin K. Towards a standardised brief outcome measure: psychometric properties and utility of the CORE-OM. Br J Psychiatry. 2002 Jan;180:51-60. doi: 10.1192/bjp.180.1.51. PMID 11772852
- [Background] Feixas, G., Alabèrnia-Segura, M. & García-Gutiérrez, A. (July, 2022). Using Virtual Reality to investigate self-identity: A case illustration of EYME-Explore Your Meanings. Paper presented in the panel Applied Personality Psychology (Chair: M. Cordero). 20th European Conference of Personality. Madrid
- [Background] Feixas, G., Carulla-Flix, A. et al (2023). Adaptación al español y propiedades psicométricas de la Escala de Autoevaluación de la Metacognición. Manuscript in preparation.
- [Background] Feixas, G. y Cornejo, J. M. (1996). Manual de la técnica de rejilla mediante el programa RECORD ver. 2.0. Barcelona: Paidós.
- [Background] Feixas, G., Fernández-Espejo, M., et al (2023). Adaptación al español y propiedades psicométricas de la Escala de Claridad de Autoconcepto. Manuscript in preparation..
- [Background] Feixas, G., Geldschläger, H., Carmona, M. y Garzón, B. (2002). Sistema de categorías de contenido para codificar constructos personales. Revista de Psicología General y Aplicada, 55, 337-348.
- [Background] Feixas, G., Pucurull, O., Roca, C., Paz, C., García-Grau, E., Bados, A. (2012). Escala de Satisfacción con el tratamiento recibido (CRES-4): La versión en español. Revista de Psicoterapia, 89(23), 51-58.
- [Background] Fonagy P, Luyten P, Moulton-Perkins A, Lee YW, Warren F, Howard S, Ghinai R, Fearon P, Lowyck B. Development and Validation of a Self-Report Measure of Mentalizing: The Reflective Functioning Questionnaire. PLoS One. 2016 Jul 8;11(7):e0158678. doi: 10.1371/journal.pone.0158678. eCollection 2016. PMID 27392018
- [Background] Fransella, F., Bell, R. y Bannister, D. (2004). A Manual for Repertory Grid Technique (2nd. ed.). Wiley.
- [Background] Garcia-Gutierrez, A. y Feixas, G. (2018). GRIDCOR: A Repertory Grid Analysis Tool (Version 6.0) [Web application]. Retrieved from http://www.repertorygrid.net/en
- [Background] Katznelson H. Reflective functioning: a review. Clin Psychol Rev. 2014 Mar;34(2):107-17. doi: 10.1016/j.cpr.2013.12.003. Epub 2013 Dec 29. PMID 24486522
- [Background] Kelly, G. A. (1955). The Psychology of Personal Constructs (2 vols). Norton.
- [Background] Lang TA, Altman DG. Basic statistical reporting for articles published in biomedical journals: the "Statistical Analyses and Methods in the Published Literature" or the SAMPL Guidelines. Int J Nurs Stud. 2015 Jan;52(1):5-9. doi: 10.1016/j.ijnurstu.2014.09.006. Epub 2014 Sep 28. No abstract available. PMID 25441757
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Martin-Albo J, Nuniez JL, Navarro JG, Grijalvo F. The Rosenberg Self-Esteem Scale: translation and validation in university students. Span J Psychol. 2007 Nov;10(2):458-67. doi: 10.1017/s1138741600006727. PMID 17992972
- [Background] Morejón, A. J. V., García-Bóveda, R. J., y Jiménez, R. V. (2004). Escala de autoestima de Rosenberg: fiabilidad y validez en población clínica española. Apuntes de Psicología, 22(2), 247-255.
- [Background] Pedone, R., Semerari, A., Riccardi, I., Procacci, M., Nicolò, G., & Carcione, A. (2017). Development of a self-report measure of metacognition: The metacognition self-assessment scale (MSAS). Instrument description and factor structure. Clinical Neuropsychiatry, 14(3), 185-194.
- [Background] Rosenberg, M. (1965). Society and the adolescent self-image. Princeton University Press.
- [Background] Ruiz-Parra E, Manzano-Garcia G, Mediavilla R, Rodriguez-Vega B, Lahera G, Moreno-Perez AI, Torres-Cantero AM, Rodado-Martinez J, Bilbao A, Gonzalez-Torres MA. The Spanish version of the reflective functioning questionnaire: Validity data in the general population and individuals with personality disorders. PLoS One. 2023 Apr 6;18(4):e0274378. doi: 10.1371/journal.pone.0274378. eCollection 2023. PMID 37023214
- [Background] Trujillo A, Feixas G, Bados A, Garcia-Grau E, Salla M, Medina JC, Montesano A, Soriano J, Medeiros-Ferreira L, Canete J, Corbella S, Grau A, Lana F, Evans C. Psychometric properties of the Spanish version of the Clinical Outcomes in Routine Evaluation - Outcome Measure. Neuropsychiatr Dis Treat. 2016 Jun 21;12:1457-66. doi: 10.2147/NDT.S103079. eCollection 2016. PMID 27382288
- [Background] Neimeyer, R. A. (1993). Constructivist approaches to the measurement of meaning (pp. 58-103). In G. J. Neimeyer (Ed) Constructivist Assessment: A Casebook. Sage.